CLINICAL TRIAL: NCT05505786
Title: The Effects of Increased vs. Traditional Squat Stance Width on Performance Indices in Elite Rugby League Players; an 8-week Pre-season Randomized Control Intervention
Brief Title: The Effects of Increased vs. Traditional Squat Stance Width on Performance Indices in Elite Rugby League Players
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Central Lancashire (Other)
Responsible Party: Principal Investigator, Jonathan Sinclair, Professor, University of Central Lancashire
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: Squat stance width
Record Dates: First submitted 2022-08-16; First posted 2022-08-18 (Actual); Last update posted 2022-09-06 (Actual); Status verified 2022-08

CONDITIONS: Sports Performance

STUDY DESIGN:
Intervention Model Description: Stratified to include similar number of forward and backs in each arm.
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Normal stance width (Active Comparator): Those assigned to this group will complete their pre-season training as normal i.e. when performing their squat exercises they will do so using their habitual (self-selected) stance width.
  Interventions: Behavioral: Normal stance width
- Wide stance width (Experimental): Those assigned to this (i.e. experimental) group will also complete their pre-season training as normal, the only exception will be that when performing their squat exercises they will increase their stance width by 20% compared to their self-selected stance width.
  Interventions: Behavioral: Wide stance width

INTERVENTIONS:
Behavioral: Normal stance width — Normal self-selected stance width when performing squat exercises.
  Arms: Normal stance width
Behavioral: Wide stance width — Increased stance with (by 20% over their own self-selected stance width) when performing squat exercises.
  Arms: Wide stance width

SUMMARY:
The back squat is a commonly utilized resistance training exercise for the promotion of both performance and musculoskeletal health. There are a range of manipulations that can be made to the setup of this resistance exercise, with once such adaptation being the stance width when performing the exercise. This intervention aims to explore the effects of increasing the stance with on performance indices in elite rugby league players.

ELIGIBILITY:
Inclusion Criteria:

* Rugby league player contracted to a professional Super League team
* 5-years minimum of back squat experience
* Male
* Injury free for 6-months

Exclusion Criteria:

* Female
* Any injury at baseline
* Any international matches played during the between season break

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2022-04-01 (Actual)

PRIMARY OUTCOMES:
505 agility test | Baseline
  Test of 180 degree turning ability, measured using timing gates.
505 agility test | 8-weeks
  Test of 180 degree turning ability, measured using timing gates.

SECONDARY OUTCOMES:
Body mass | Baseline
  Body mass using a weighing scale.
Body mass | 8-weeks
  Body mass using a weighing scale.
Sum of skinfold thickness | Baseline
  Skinfold thicknesses measured using callipers at eight sites according to the International Society for the Advancement of Kinanthropometry (ISAK) restricted profile (triceps, subscapular, biceps, iliac crest, supraspinal, abdominal, mid-thigh, and medial calf)
Sum of skinfold thickness | 8-weeks
  Skinfold thicknesses measured using callipers at eight sites according to the International Society for the Advancement of Kinanthropometry (ISAK) restricted profile (triceps, subscapular, biceps, iliac crest, supraspinal, abdominal, mid-thigh, and medial calf)
Three repetition maximum squat strength | Baseline
  The maximum squat weight that can be lifted for a total of three repetitions
Three repetition maximum squat strength | 8-weeks
  The maximum squat weight that can be lifted for a total of three repetitions
Counter movement jump height | Baseline
  The maximum height that can be jumped vertically, measured using a jump mat.
Counter movement jump height | 8-weeks
  The maximum height that can be jumped vertically, measured using a jump mat.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Central Lancashire, Preston, Lancashire, United Kingdom

IPD SHARING:
Plan to Share IPD: No